CLINICAL TRIAL: NCT03072511
Title: Pilot Trial of a Smoking Cessation Intervention Informed by Construal Level Theory
Brief Title: Smoking Cessation Intervention
Acronym: SPOTLIGHT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: PI is relocating to another institution.
Sponsor: University of Florida (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB201601307 - N; K02DA034767 (NIH)
Record Dates: First submitted 2017-03-01; First posted 2017-03-07 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Spotlight on Smoke-Free Living (Experimental): Treatment will include a 1.5-hour intervention session combined with daily text-messaging for up to 1 week pre-quit and 4 weeks post-quit. The intervention includes: mindful breathing, visualization, and identification and thinking about goals and priorities inconsistent with smoking. During the text-messaging phase, elements of the intervention discussed during the in-person session will be reinforced. Participants will be provided transdermal nicotine patches (TNP). TNP are a safe and effective approach to nicotine replacement when an individual attempts to stop smoking and are safe for use without prescription. Participants will begin the regimen on the scheduled quit date with an initial dose of 21 mg (4 weeks), followed by 14 mg (2 weeks), and 7 mg (2 weeks). Alterations to dosing will be allowed when appropriate and consistent with manufacturer's recommendations. While TNP will be offered to all participants, they can decline or discontinue use of TNP at any time.
  Interventions: Behavioral: Spotlight on Smoke-Free Living: Mindsets and Decisions; Drug: Transdermal Nicotine Patch
- Standard Informational Treatment (Active Comparator): Standard informational treatment is based on conventional, information-based smoking cessation approaches commonly found in public health settings. This will include the following information: prevalence/incidence of cigarette smoking and negative health outcomes associated with cigarette smoking (e.g., cancer, respiratory disease, complications), other health consequences resulting from diseases associated with cigarette smoking, personal/financial/social consequences of cigarette smoking. During the text-messaging phase, information about the consequences of smoking discussed during the in-person session will be reiterated. As with the experimental condition, participants will be provided with 8-weeks TNP.
  Interventions: Drug: Transdermal Nicotine Patch

INTERVENTIONS:
Behavioral: Spotlight on Smoke-Free Living: Mindsets and Decisions — Intervention will consist of elements to help quit smoking. All intervention elements will be informed by Construal Level Theory.
  Other Names: SPOTLIGHT
  Arms: Spotlight on Smoke-Free Living
Drug: Transdermal Nicotine Patch — TNP serve as nicotine replacement for individuals who are attempting to stop smoking. They are safe for use and dosing will be determined for each participant based off of manufacturer's recommendations.
  Other Names: TNP

SUMMARY:
Cigarette smoking is the leading cause of preventable mortality in the United States, yet less than 10% of smokers making a serious quit attempt remain abstinent from cigarettes 1 year later, and outcomes from gold-standard behavioral interventions leave much room for improvement. As such, in the context of a Stage-I randomized controlled trial (RCT), this study will examine (1) treatment characteristics and delivery, treatment integrity, dropout, and acceptability, (2) smoking outcomes such as lapse, relapse, and abstinence measures, and (3) changes decision-making that result from a novel intervention informed by behavioral analysis and social cognition.

DETAILED DESCRIPTION:
Cigarette smoking is the leading cause of preventable mortality in the United States, implicated in countless health consequences, and significant economic and societal costs. Less than 10% of smokers making a serious quit attempt remain abstinent from cigarettes 1 year later, and outcomes from gold-standard behavioral interventions leave much room for improvement. Thus the development of new interventions and improvements to existing interventions is imperative. Behavioral interventions for smoking cessation have insufficiently integrated the findings from basic research on decision-making processes. Thus, there is extensive laboratory-based research indicating the potential for laboratory-based manipulations that affect decision making relevant for smoking, the examination of a coherent intervention that capitalizes on this knowledge is limited. The proposed research is the first step toward synthesizing insights from the research domains of addiction, behavioral analysis, and social cognition into a cohesive formulation with potential impact on smoking cessation. Specifically, the research targets impulsive decision making associated with cigarette smoking and relapse by incorporating the influential Construal Level Theory.

ELIGIBILITY:
Inclusion Criteria:

* Current cigarette smoker (verified with an expired carbon monoxide level of at least 4 ppm of expired air),
* At least 18 years of age,
* With a desire to quit smoking in the next month (at least 5 on a 10-point scale).

Exclusion Criteria:

* Pregnancy,
* Having uncontrolled serious psychiatric or medical illnesses,
* Having recent suicide attempts or ideation,
* Meeting contraindications for use of nicotine replacement products,
* Taking pharmocotherapy for smoking cessation treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-12-13 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
7-day smoking point prevalence | 13 weeks
  Timeline Follow-Back: assesses smoking patterns through daily logs of smoking tendencies, use of nicotine patches, and attempts to quit.
Delay Discounting | 13 weeks
  Delay Discounting Task: a binary choice procedure where two hypothetical money rewards will be presented at specified delays.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Yi, Ph.D., Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided